CLINICAL TRIAL: NCT00001466
Title: Clinical and Molecular Manifestations of Six Categories of Genetic Disorders
Brief Title: Study of Clinical and Molecular Manifestations of Genetic Disorders
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950010; 95-HG-0010
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-09

CONDITIONS: Hereditary Diseases
Keywords: Clinical Genetics; Etiology; Medical Screening; Prognosis; Genetic Disorders
MeSH Terms: conditions — Genetic Diseases, Inborn

SUMMARY:
This study will investigate the cause and natural history (medical problems that appear over time) of certain genetic disorders. It will also try to locate the abnormal genes responsible for these conditions and eventually develop tests to predict who is likely to be affected and to what degree.

Patients with known or suspected genetic disorders in certain categories, such as those involving chromosomal or metabolic abnormalities, immune system or blood disorders, abnormal growth, benign tumors, and others may be eligible for this study. Participants will be interviewed by specialists in genetics about their condition and family history. They may also be asked to have a physical examination and certain tests needed for study of the specific individual's condition. These may include collection of blood samples (up to 3 tablespoons); imaging studies, such as computerized tomography (CT), magnetic resonance imaging (MRI), ultrasound and echocardiography; skin biopsy (removal of a small sample of skin tissue under local anesthetic), and other procedures. DNA testing may reveal the genetic abnormality responsible for the disorder. Participants who so wish will have an opportunity to talk with experts about the health implications of the test results.

This study may provide information that will lead to improved treatment or management of these inherited disorders, as well as more effective genetic counseling for families.

DETAILED DESCRIPTION:
Individuals and their families affected by disorders with a potentially genetic basis within six broad categories will be evaluated over time to characterize the natural and clinical history of various specific disorders. Medical and laboratory evaluations will be completed to identify areas of management concern that have not been previously described. Further protocols will be developed addressing specific disorders once a number of affected individuals have been investigated and is sufficient to query various aspects of those disorders. Issues for both diagnosis and medical management of those affected with certain genetic disorders will be collated and addressed within a national consensus conference format. In addition, phenotype to genotype correlation will be established to further understanding of specific molecular alterations on phenotypic expression. This broad-based protocol will also facilitate the training of fellows in medical genetics, graduate and post graduate training in genetics and genetic counseling.

ELIGIBILITY:
Patients and their families with known or suspected genetic disorders within the following categories will be recruited:

Hereditary connective tissue disorders;

Phacomatoses;

Chromosomal disorders;

Dysmorphic syndromes;

Neuromuscular or neurological disorders;

Inherited immunological and hematologic disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200
Dates: Start 1994-10; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States